CLINICAL TRIAL: NCT06885294
Title: Impact of Physiotherapy Combined to Hypnosis on Superior Limb Functional Capacities of AVC Patients
Brief Title: Physiotherapy/hypnosis for AVC Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-306
Record Dates: First submitted 2024-04-08; First posted 2025-03-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Hypnosis, Stroke, physiotherapy
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 receiving physiotherapy only (Experimental): Stroke patients will receive physiotherapy of upper limbs
  Interventions: Behavioral: Physiotherapy
- Group 2 receiving combined physiotherapy and hypnosis (Experimental): Stroke patients will receive physiotherapy of upper limbs under hypnosis
  Interventions: Behavioral: Physiotherapy and Hypnosis
- Waitlist group 3 receiving delayed combined physiotherapy and hypnosis (Experimental): Stroke patients will receive physiotherapy of upper limbs under hypnosis one month after the other groups
  Interventions: Behavioral: Control group Physiotherapy and Hypnosis

INTERVENTIONS:
Behavioral: Physiotherapy — Stroke patients will be randomly assigned to join one of the three groups. The first group will undergo a pre-treatment evaluation, receive 6 sessions of physiotherapy (2 sessions per week, approximately 20-30 minutes each), and undergo a post-treatment evaluation after 1 month. After another month without any treatment, they will undergo a third and final assessment. All evaluations will last approximately 1 hour.
  Arms: Group 1 receiving physiotherapy only
Behavioral: Physiotherapy and Hypnosis — Stroke patients will be randomly assigned to join one of the three groups. The second group will undergo a pre-treatment evaluation, receive 6 sessions of physiotherapy combined with hypnosis (2 sessions per week, approximately 20-30 minutes each), and undergo a post-treatment evaluation after 1 month. Patients will continue their standard physiotherapy care during these 4 weeks. After another month without any treatment, they will undergo a third and final assessment. All evaluations will last approximately 1 hour.
  Arms: Group 2 receiving combined physiotherapy and hypnosis
Behavioral: Control group Physiotherapy and Hypnosis — The control group will be assessed initially and then after 4 weeks. After the second assessment, they will receive 6 sessions of physiotherapy combined with hypnosis (2 sessions per week, approximately 20-30 minutes each), and undergo a post-treatment evaluation after 1 month. All evaluation sessions will last approximately 1 hour.
  Arms: Waitlist group 3 receiving delayed combined physiotherapy and hypnosis

SUMMARY:
Impact of physical therapy with hypnosis on the functional capacity of the upper limb in stroked patients.

DETAILED DESCRIPTION:
The cerebrovascular accident (CVA) is a pathology generating many disabled people. Physiotherapy is one of the usual rehabilitation techniques for a patient with sequelae of ischemia or cerebral hemorrhage. Combined with another therapeutic approach, hypnosis, it could increase the patient's motor performance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years old
* Having experienced a stroke more than 3 months ago
* Understanding and proficient in the French language
* Having a functional capacity deficit in at least one of the two upper limbs
* Being able to independently travel to the Yerne medical center for necessary study appointments.

Exclusion Criteria:

* Being under 18 or over 80 years old
* Having a history of upper limb injuries (fractures, prosthetics, etc.)
* Having Wernicke's aphasia (language comprehension disorder)
* Having frontal lobe syndrome
* Undergoing chemotherapy
* Having respiratory disorders (respiratory failure of more than 70%) or receiving oxygen therapy
* Having epilepsy
* Having dementia
* Having untreated hearing impairments
* Being diagnosed with schizophrenia or paranoïa
* Experiencing significant concentration difficulties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of joint ranges of motion | 8 weeks
  Measurement of shoulder (flexion, extension, abduction, internal rotation, external rotation), elbow (flexion, extension), wrist (flexion, extension)
assessment of spasticity | 8 weeks
  Measurement of muscle activation on Ashworth scale (extension and flexion of shoulder, elbow, wrist, fingers, thumb) => 0%-100% (a higher score means a worse outcome)
functional tests for the upper limb | 8 weeks
  Stroke Upper Limb Capacity Scale (SULCS) => 0%-100% (a higher score means a better outcome)
  * using one forearm as support while sitting
  * wedging an object between the chest and the upper part of the affected limb
  * sliding an object across a table while sitting
  * partially unscrewing a lid
  * taking a glass of water and drinking it
  * grabbing a tennis ball presented at a certain height
  * coming one's hair with the affected upper limb
  * buttoning
  * writing
scales for assessing disability and functional independence | 8 weeks
  Functional Independence Measure (FIM) from complete dependence to independence => 0%-100% (a higher score means a better outcome)
  * personal care
  * sphincter control
  * mobility, transfers
  * locomotion
  * communication
  * awareness of the external world
evaluation of muscle strength | 8 weeks
  Measurement of pathological upper limb strength on MRC scale by group/time/joint/movement => 0%-100% (a higher score means a better outcome)
  * Shoulder Flexion Strength
  * Shoulder Extension Strength
  * Shoulder Abduction Strength
  * Shoulder Internal Rotation Strength
  * Shoulder External Rotation Strength
  * Elbow Flexion Strength
  * Elbow Extension Strength
  * Wrist Flexion Strength
  * Wrist Extension Strength
  * Finger Flexion Strength
  * Finger Extension Strength
  * Thumb Flexion Strength
  * Thumb Extension Strength
Box and Block Test (BBT) | 8 weeks
  Measurement of manual dexterity and motor skills by moving blocks into box comparing healthy upper limb with pathological upper limb => 0%-100% (a higher score means a better outcome)
Modified Rankin Scale (mRS) | 8 weeks
  Measurement of degree of disability => 0%-100% (a higher score means a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Vanhaudenhuyse, PhD, Study Director — University of Liege
Locations (1):
- GIGA Science and Perception Research Group CHU Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No